CLINICAL TRIAL: NCT07034339
Title: Construction and Clinical Application of the Immune Map of Pancreatic Cancer Evolution
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Qi Zhang, Professor, First Affiliated Hospital of Zhejiang University
Other Study IDs: IDPEPDAC
Record Dates: First submitted 2025-06-15; First posted 2025-06-24 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Immune Evasion, Tumor; Pancreas Cancer
MeSH Terms: conditions — Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Conventional treatment queue
- Dynamic follow-up queue
- Neoadjuvant therapy queue

SUMMARY:
The intricate interplay between systemic immunity and tumors profoundly influences not only the onset and progression of tumors but also serves as a crucial window into understanding tumor evolution and treatment status. This project aims to establish a large, multi-center pancreatic cancer cohort and a standardized clinical sample repository, capturing multimodal immunity big data on pancreatic cancer occurrence, progression, and treatment response across the spatial dimension of "peripheral versus local" and the temporal dimension of "tumor evolution/pre- and post-treatment." By integrating patient imaging and clinical information, the investigators will develop a technical platform for intelligent extraction and fusion analysis of cross-scale, multimodal data, thereby mapping the immunity landscape of pancreatic cancer evolution, identifying characteristic changes in immunity parameters, and devising an AI model for early pancreatic cancer diagnosis with high accuracy and robust generalization capabilities, while also exploring the model's interpretability. Additionally, the investigators will focus on specific immune cell subsets associated with pancreatic cancer evolution and treatment response, elucidating their roles and mechanisms in the occurrence, development, and drug resistance of pancreatic cancer. This project will establish a high-quality, standardized, and shareable pancreatic cancer immunity sample and data repository, refine the framework for multi-dimensional immunity data fusion and analysis, and create a time-space atlas of local and systemic immunity in pancreatic cancer. This will facilitate a deeper understanding of the dynamics of systemic and local immunity in early-stage pancreatic cancer and at various stages of its evolution, offering novel insights and approaches for the diagnosis and treatment of pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals without benign or malignant liver, gallbladder, and pancreas diseases
* Primary PDAC
* Patients with benign pancreatic tumors
* IPMN patients diagnosed by pathology/imaging

Exclusion Criteria:

* Having autoimmune diseases
* Accompanied by other malignant tumors
* History of tumor treatment (except thyroid cancer and breast cancer, cured for more than 5 years)
* Acute infection
* History of blood transfusion within the past 6 months, or use of drugs that affect peripheral blood components such as recombinant human erythropoietin and interleukin within 2 weeks
* Organ decompensation dysfunction
* Immunodeficiency syndrome
* Hematological precancerous lesions
* Accept immunosuppressive therapy
* Diagnosed coagulation disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with pancreatic cancer, benign diseases, and healthy
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pancreatic tumor resection | 3 years
  Number of participants with pancreatic cancer

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China